CLINICAL TRIAL: NCT04882020
Title: Inflammation and Neurocognitive Damage Markers in Elderly People With Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0529
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Obstructive Sleep Apnea; Sleep Apnea; Apnea, Obstructive; Obstructive Sleep Apnea Syndrome; Inflammation; Inflammatory Response; Neurocognitive Disorders; Neurodegenerative Diseases
Keywords: Obstructive Sleep Apnea; Inflammation; Neurocognitive Damage
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Inflammation; Neurocognitive Disorders; Neurodegenerative Diseases | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma stored at -80ºC in Molecular and Protein Analysis Unit (UAMP) of Hospital de Clínicas de Porto Alegre, Rio Grande do Sul, Brazil.
  All rates who will not suffer any type of intervention in the studies of the MEDIDAS cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AHI ≤ 5: Individuals aged 65 to 80; both sexes; Informed Consent Form with prior signature for participation in the MEDIDAS cohort study; previous performance of ambulatory polysomnography with adequate technical quality and AHI ≤ 5 events / hour; prior blood collection between 7-9 am and questionnaires.
  Interventions: Diagnostic Test: cortisol, BDNF, s100B, IL-1B, IL-6, IL-10, TNF-alpha
- AHI ≥ 30: Individuals aged 65 to 80; both sexes; Informed Consent Form with prior signature for participation in the MEDIDAS cohort study; previous performance of ambulatory polysomnography with adequate technical quality and AHI ≥ 30 events / hour; prior blood collection between 7-9 am and questionnaires.
  Interventions: Diagnostic Test: cortisol, BDNF, s100B, IL-1B, IL-6, IL-10, TNF-alpha

INTERVENTIONS:
Diagnostic Test: cortisol, BDNF, s100B, IL-1B, IL-6, IL-10, TNF-alpha — compare both groups and evaluate the severity of obstructive sleep apnea modulates serum levels of inflammatory and neurocognitive markers in elederly.
  Other Names: polysomnography; Beck Depression Inventory; Mini-Mental State Examination (MMSE); WHOQOL-OLD questionnaire

SUMMARY:
The aging process tends to promote an overall increase in inflammation compromising the immunologic system regulation, sleep/wakefulness pattern, and neurocognitive performance. In elders, there is an increase in repetitive arousals during sleep, secondary to breathing interruption by pharynx collapse, generating a transient reduction in oxygen delivery to the brain known as obstructive sleep apnea. This lack in oxygen supply results in an inflammatory process producing brain damage. Some substances present in the blood seem to be associated to neurocognitive damage, like S100β protein, cortisol, interleukin 1-β,6 and TNF-α. In the other way, a substance called brain-derived neurotrophic factor (BDNF) enhances cognitive function, and memory consolidation improvement.

DETAILED DESCRIPTION:
An intermittent hypoxia in obstructive sleep apnea induces the production of reactive oxygen species (ROS), oxidative damage and inflammation generating pro-inflammatory cytokines, reactive gliosis and neuronal damage. The increase in oxidative damage seems to be associated to age, contributing to the progress of neurodegeneration. Transient hypoxemia leads to autonomic excitation causing hyperactivity of the sympathetic nervous system (SNS), and activation of the hypothalamic-pituitary-adrenal (HPA) axis, causing immunological changes and increased risk of damage to mental functions. Night awakenings caused by OSA are associated with changes on the HPA axis, resulting in increased serum cortisol levels. The fluctuation in serum cortisol levels at night is intrinsically related to sleep, and increases with advancing age. BDNF is responsible for increasing the growth of neurites, and synaptogenesis, preventing programmed cell death in adults, and is involved in stress responses on the HPA axis. Low BDNF levels are associated to cognitive impairment, less memory consolidation, depression, and OSA. There is a positive correlation between levels of BDNF and cortisol related to physiological regulation of brain activities. The increase in oxidative damage caused by intermittent hypoxia during obstructive sleep apnea increases serum levels of the s100β protein promoting reactive gliosis or astrogliosis being associated to depression in the elderly. Obstructive sleep apnea syndrome is associated with development of cardiovascular and neurological diseases by activating pro-inflammatory pathways. However, in elderly individuals, regardless of other specific pathologies, they already have a pro-inflammatory state secondary to loss of regulation of the immune system.

ELIGIBILITY:
Inclusion criteria:

* Individuals aged 65 to 80;
* both sexes;
* free and informed consent form previously signed for participation in the MEDIDAS cohort study;
* previous performance of outpatient polysomnography with adequate technical quality
* AHI ≤ 5 or ≥ 30 events/hour;
* previous blood collection between 7-9 am; questionnaires.

Exclusion criteria:

* Have had treatment for sleep apnea;
* suffer from rheumatic or chronic diseases such as diabetes mellitus, heart failure, coronary artery disease, chronic renal failure or nephropathy (creatinine> 1.8 mg / dL), liver disease, history of stroke, aortic aneurysm, marked elevation in blood arterial pressure (> 180/110 mmHg), assessed by 24-hour ambulatory blood pressure monitoring (ABPM);
* cognitive deficit verified in the Mini Mental State Examination;
* diagnosis of Alzheimer's and Parkinson's.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: A sample will be composed from the database and the biorepository of volunteers participating in the MEDIDAS cohort study. The database was stored in the Non-Invasive Methods Unit (UMNI) and the biorepository of blood aliquots initiated at -80ºC in the Molecular and Protein Analysis Unit (UAMP) in Hospital de Clínicas de Porto Alegre, Brazil. All data and aliquots will not suffer any type of intervention in the studies of the MEDIDAS cohort.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-11 (Estimated)

PRIMARY OUTCOMES:
Serum level of Brain derived neurotrophic factor | Baseline
  Serum of brain-derived neurotrophic factor will be analyzed in the plasma of elderly volunteers using the Sandwich ELISA method.

SECONDARY OUTCOMES:
Serum level of s100B protein | Baseline
  Serum of s100B protein will be analyzed in plasma in elderly volunteers using ELISA method.
Inflammatory markers | Baseline
  The serum levels of cytokines (IL-1b, IL-6, IL-10 and TNF-alpha) will be analyzed in the plasma of elderly volunteers. The serum level of cytokines using a unit multiplex assay in pg/mL.
Serum Cortisol levels | Baseline
  Serum cortisol levels will be analyzed in the plasma of elderly volunteers. The serum level of cortisol will be quantified by chemiluminescence microparticle immunoassay (CMIA) with reference values for blood collection performed in the morning shift from 3.7 to 19.4 ug / dL.
Neurocognitive Damage | Baseline
  Neurocognitive damage will be measured by the Mini Mental State Examination adapted for the Brazilian population. The maximum score for this scale is 30 points, indicating better cognitive performance. A score of 0-9 points indicates severe cognitive loss; 10-20 points of moderate cognitive loss; 21-26 points mild cognitive loss, 27-30 points without cognitive loss.
Depression | Baseline
  Depression will be measured by the Beck Depression Inventory. A score of 0-9 points indicates that the individual is not depressed; 10-18 points mild depression; 19-29 points moderate depression; 30-36 points severe depression.
Quality of life Score | Baseline
  Quality of life will be measured using the World Health Organization's Quality of Life questionnaire, which has assessments in the domains: physical, psychological, social relations and the environment. The evaluation of each domain is expressed as a percentage, where the higher the result (100%) indicates the better quality of life in the respective domain. The general quality of life is given by the average of the scores of the four domains, whose scores vary from 0 to 5 points. 1-2.9 points the quality of life needs to improve; 3-3.9 regular quality of life; 4-4.9 good quality of life; 5 very good quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ruy S Moraes Filho, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No